CLINICAL TRIAL: NCT01825005
Title: Predicting Outcome in Cervix Carcinoma: a Prospective Study
Acronym: POCER
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 12-4-008
Record Dates: First submitted 2013-03-12; First posted 2013-04-05 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- group 1:surgery: treatment = surgery only
- group 2: radiotherapy: treatment = radiotherapy only
- group 3: RT and CT, and/or hyperthermia: treatment= radiotherapy combined with chemotherapy and/or hyperthermia
- group 4: stage IVb , any treatment: cervical cancer stage IV b, treatment = any systemic or radiation therapy and supportive care

SUMMARY:
The main aim is to validate and improve the predictive model for survival and toxicity in patients with cervical cancer through multicentric prospective data collection. The data contain information on patient, tumor and treatment characteristics. For this study, additional health related QOL scores will be assessed using the EORTC Quality of Life Questionair-CX24 and C30. The long term aim, beyond this specific study, is to build a Decision Support System based on the predictive model validated in this study.

ELIGIBILITY:
Inclusion Criteria:

* histological or cytological proven cervical cancer
* informed consent according to national rules

Exclusion Criteria:

* no histological or cytological proven cervical cancer
* no informed consent according to national rules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with cervical cancer can be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2013-02; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
five-year overall survival rate | 5 years after treatment
  assessment of the overall survival 5 years after treatment

SECONDARY OUTCOMES:
three-year distant disease free survival | 3 years
  assessment of distant disease free survival, 3 years after treatment
three-year local disease free survival | 3 years
  assessment of local disease free survival, 3 year after treatment
five-year distant disease free survival | 5 years
  assessment of distant disease free survival,5 years after treatment
five-year local disease free survival | 5 years
  assessment of local disease free survival, 5 years after treatment
number of participants with early adverse events as a measure of safety and tolerability | 2 months
number of participants with late adverse events as a measure of safety and tolerability | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: P Lambin, Prof, Principal Investigator — Maastricht University hospital, dep of radiotherapy (Maastro clinic)
Locations (2):
- Maastricht University Hospital, Maastricht, Netherlands
- Bloemfontein medicross, Bloemfontein, Free State, South Africa